CLINICAL TRIAL: NCT06527131
Title: Pulsed Electromagnetic Field Stimulation and Charcot Foot Ulcer: a Randomized Controlled Trial
Brief Title: Pulsed Electromagnetic Field Stimulation and Charcot Foot Ulcer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Norhan Mohamed Eltayeb, Bachelor's degree, MSc candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005154
Record Dates: First submitted 2024-07-15; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Charcot Foot Ulcer
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation; Vancomycin

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Study group) (Experimental): PEMF group who recieves pulsed electromagnetic field therapy and electrical stimulation
  Interventions: Device: pulsed electromagnetic field therapy; Device: Transcutanous electrical nerve stimulation
- Group B(control group) (Active Comparator): who recieves standard wound care , electrical stimulation and medical treatment
  Interventions: Device: Transcutanous electrical nerve stimulation; Drug: Vancomycin

INTERVENTIONS:
Device: pulsed electromagnetic field therapy — PEMF is regarded as an efficient physical therapy method that has been utilized clinically to treat a variety of orthopedic conditions, including delayed union and nonunion of fractures. According to studies, PEMF has been authorized for its biological effects, which include the mineralization of bone matrix, osteogenic differentiation of mesenchymal stem cells, and osteoblast proliferation
  Other Names: PEMF
  Arms: Group A (Study group)
Device: Transcutanous electrical nerve stimulation — Electrical stimulation consider a safe and cost-effective method for pain management. It has no side effects and few contraindication in addition to no drug interaction . According to studies ,electrical stimulation decreases pain through reducing central transmission of pain signals because of nociceptive inhibition at the presynaptic level in the dorsal horn.
  Other Names: TENS
Drug: Vancomycin — medical antibiotics
  Arms: Group B(control group)

SUMMARY:
thirty-four patients with charcot foot ulcer will be included, their ages will be ranged from 50 to 70 years old and randomly distributed into two equal groups : study group includes 17 patients who will recieve pulsed electromagnetic field and electrical stimulation three days per week for three months .

control group includes 17 patients who will recieve electrical stimulation , standard wound care and medical treatment

ELIGIBILITY:
Inclusion Criteria:

* age ranges between 50 and 70 years old male and female patients all patients with charcot foot ulcer

Exclusion Criteria:

* presence of malignancy hypotensive patients pregnancy immunological and rheumatological disorders

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
rate of bone healing | Baseline and three months
  asses rate of bone healing through plain x-ray after six weeks then after twelve weeks from initiation of treatment

SECONDARY OUTCOMES:
ulcrer healing | baseline and three months
  asses wound surface area through wound surface area Tracing pre treatment ,after six weeks and after twelve weeks from initiation of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Therapy Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided